CLINICAL TRIAL: NCT03153046
Title: Effects of Modulating the Immune System With Prebiotics on Cognition and Weight in Patients With Psychosis
Brief Title: The Effects of Prebiotics on Cognitive Functioning and Weight Gain in Psychosis
Acronym: Prepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Clasado Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 12302
Record Dates: First submitted 2017-05-02; First posted 2017-05-15 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-05

CONDITIONS: Schizophrenia
Keywords: prebiotics; cognitive impairment; weight gain
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Weight Gain | interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Intervention Model Description: 24 week cross-over at 12 week involving preiotics and maltodextrin
Who Masked: Participant, Investigator
Masking Description: Blinding of compounds will be provided by Clasado Ltd., the company supplying the prebiotics and maltodextrin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotics (Experimental): 12 week ingestion of prebiotics, Bimuno galacto-oligosaccharide (B-GOS).
  Interventions: Dietary Supplement: prebiotics
- Maltodextrin (Placebo Comparator): 12 week ingestion of maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: prebiotics — Bimuno (BGOS): The active supplement of the food supplement (Bimuno) used in this study is called galacto-oliogosaccharides (Bimuno®, BGOS). BGOS is a compound metabolised by specific bifidobacteria, which are beneficial bacteria, in our colon. Bimuno (2.3 calories) is composed by the following ingredients per gram of Bimuno: 0.96g dry matter; <01g Fat; <0.06g Protein; 0.821g GOS; 0.119g Lactose; 0.0331g Glucose and 0.0029g Galactose. Bimuno is tasteless. Bimuno will be supplied in coded sachets (3.5g) for dispensing by parents. Each participant will be required to consume 1 sachet daily during breakfast, by mixing it with food or in a drink.
  Other Names: Bimuno® galacto-oliogosaccharides (BGOS)
  Arms: Prebiotics
Dietary Supplement: Maltodextrin — Maltodextrin is a polysaccharide in powder form, which grows most bacteria in the gut, and not specifically the beneficial bifidobacteria. The placebo will also be provided in daily coded sachets (3.5g) for dispensing by parents. Each participant will be required to consume 1 sachet daily during breakfast, by mixing it with food or in a drink. This placebo has been used in previous studies, in which Bimuno was used as the active intervention. The placebo will be similar in taste and colour to the active intervention.
  Arms: Maltodextrin

SUMMARY:
The investigators propose a maltodextrin-controlled cross over experimental medicine study that aims to examine the role of the immune system in cognitive processes and weight gain in 40 adult patients with psychosis, stable on antipsychotic medication for over 1 month. There is evidence suggesting the immune system is linked to brain function and weight gain, both parameters that has been implicated in psychosis and antipsychotic use, and may underlie some schizophrenic features. The fermentation of galacto-oligosaccharides (GOS), which are short chain carbohydrates composed mostly of galactose sugar molecules, by the intestinal microbiota has been shown to modulate the immune system and reduce the inflammatory response in both animals and humans. Since the intestinal ecosystem is highly sensitive to dietary changes, the growth of beneficial gut bacteria can be enhanced using a natural food supplement similar to GOS known as prebiotics. The study will be controlled by taking maltodextrin as a control supplement. Both prebiotics and maltodextrin are short chain sugar compounds. The study will involve asking patients to take dietary supplement for a total of 24 weeks; GOS for 12 weeks and maltodextrin for 12 weeks as a control. Participants will be randomised into groups, with half receiving maltodextrin followed by GOS, and half receiving GOS followed by maltodextrin. Participants will be assessed on cognitive function and weight gain at 3 specified time points.

DETAILED DESCRIPTION:
An 24-week maltodextrin-control cross-over experimental medicine study enrolling 40 patients with psychosis. Participants will receive a 12-week treatment with Bimuno™ GOS, as well as a 12-week maltodextrin supplement. The order of supplements that participants will receive is randomized. A washout period was considered unnecessary as maltodextrin is an inactive placebo wherein negligible effects have been shown on bifidobacteria growth, and therefore, would present with no carryover/lasting effects to mask the prebiotic effect.

Eligible patients will be invited to be screened for the study and assessed to ensure they meet inclusion/exclusion criteria. If the participant passes this initial screening stage and conditional to informed consent, he/she will then be randomized into one of the two groups. Once decided, the participant will be assessed by a research assistant using standard clinical assessments used to diagnose/evaluate cognitive deficits. A 12-week supply of sachets containing prebiotic or maltodextrin will be provided for the participant to allow participants to complete the first quarter of the study. Additional 12-week supplies of prebiotics or maltodextrin will be provided at the study follow-up. Since clozapine/olanzapine are well known antipsychotics that induce weight gain and interfere with the immune system an additional sub-analysis of those participants stable on clozapine/olanzapine will be performed, contingent on the demographics.

The study will include five sessions in total all taking place at either University Department of Psychiatry, Warneford Hospital, or a location convenient to the participant (e.g., patient home): (1) screening session, (2) baseline cognitive and blood measurements, (3) study follow up, and (4) final testing session.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18-60 years of age.
* Participant is willing and able to give informed consent for participation in the study
* Diagnosed with psychotic disorder ICD-10 (e.g., schizophrenia, schizoaffective disorder, psychosis NOS)
* Stable on psychotropic medication for >1 month with cognitive deficits (Cognitive deficits will be evaluated using the BACS test cut off score of 1.0 standard deviation below the healthy mean; those that score within the normal range i.e., within 1.0 standard deviations of the mean are not considered cognitively impaired and thus will not be included in the study)

Exclusion Criteria:

* Not considered suitable for the study by the clinical team, for whatever reason
* Current inpatient in psychiatric hospital
* Additional major medical disorders (including diseases affecting the human gastrointestinal tract and blood-borne disorders)
* Antibiotic, probiotic and/or prebiotic treatment in at least the 3 previous months
* Participants who are taking any other food supplements which, in the opinion of the Investigators, may affect the results
* Participants who have a known intolerance to lactose (self-identified)
* Any significant recent change in diet which, to the discretion of the Investigators, may affect the results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Cognitive Assessments using the BAC's Test | 1 year
  The Brief Assessment of Cognition (BAC), developed by NeuroCog. Trials, assesses five different domains of cognitive function with six tests (i.e., Verbal Memory & Learning (Verbal Memory), Working Memory (Digit Sequencing), Motor Function (Token Motor Task), Verbal Fluency (Semantic and Letter Fluency), Speed of Processing (Symbol Coding), and Executive Function (Tower of London)). Outcome measures from each test will be combined into one composite Z-Score, and transformed into a T-Score to evaluate global cognition on a standardise curve.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 1 year
  Weight in kilograms and height in meters will be measured to calculate the BMI kg/m^2 of a participant.
Waist-Hip Ratio | 1 year
  Waist and hip circumference will be measured in centimeters where the Waist-to-Hip ratio will calculated.
Circulating Inflammatory Markers | 1 year
  Collected venous blood will be spun down to isolate plasma wherein biochemical tests examining inflammatory markers including interleukin-1b, tumour necrosis factor alpha, interleukin-8 and acetate will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Lennox, MD, Principal Investigator — University of Oxford
Locations (1):
- Warneford Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kao AC, Safarikova J, Marquardt T, Mullins B, Lennox BR, Burnet PWJ. Pro-cognitive effect of a prebiotic in psychosis: A double blind placebo controlled cross-over study. Schizophr Res. 2019 Jun;208:460-461. doi: 10.1016/j.schres.2019.03.003. Epub 2019 Mar 12. No abstract available. PMID 30876680